CLINICAL TRIAL: NCT01296269
Title: Effects of Intranasal Oxytocin and Vasopressin on Social Behavior in Healthy Controls
Brief Title: Effects of Intranasal Oxytocin and Vasopressin on Social Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: David Mankuta MD, Hadassah Ein-Kerem - obstetrics and gynecology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OXTandAVP-HMO-CTIL
Record Dates: First submitted 2011-02-03; First posted 2011-02-15 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: social cognition; oxytocin; vasopressin; decision making; social decision making
MeSH Terms: conditions — Diabetes Insipidus | interventions — Oxytocin; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vasopressin (Experimental): vasopressin condition
  Interventions: Drug: Arginine Vasopressin
- oxytocin (Experimental): oxytocin condition (syntocinon)
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oxytocin — one-time intranasal administration, 24 International Units, 5 puffs for each nostril
  Other Names: syntocinon
  Arms: oxytocin
Drug: Arginine Vasopressin — one-time intranasal administration, 20 International Units, 5 puffs in each nostril
  Arms: Vasopressin
Drug: placebo — contains all the ingredients as in the oxytocin and vasopressin conditions, save for the active ingredient, one time intranasal administration, 5 puffs in each nostril
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the role of a one-time intranasal administration of the oxytocin, vasopressin, or placebo on prosocial decision making such as cooperation and altruism in a healthy population of student controls.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls

Exclusion Criteria:

* Past or present psychiatric, neurological, endocrinological or severe chronic medical illness.
* Use of medications or drugs that would interfere with study results. This includes steroids, medications for psychiatric symptoms like anxiety or depression, stimulants, and medications for high blood pressure. Participants will be asked to tell the investigators of any medications or drugs that they are taking. The investigators will consider the drug interactions with oxytocin and vasopressin prior to study, and participants will not be able to participate in the study if the drug interactions could be dangerous.
* history of drug or alcohol addiction
* Pregnancy or Nursing Status: Because of the risk to an unborn fetus or infant, women who are pregnant or nursing are excluded from this protocol. All females will have a pregnancy test performed no more than 24 hours before each drug administration and will not be able to participate if the pregnancy test is positive.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
allocations of monetary units | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Participants will make decisions regarding the allocation of monetary units between themselves and other participants. We will measure the quantity of monetary units kept for themselves vs. given to other participants

SECONDARY OUTCOMES:
mood as measured via the visual analog scale | approximately one hour and fifteen minutes after administration of oxytocin, vasopressin or placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, MD, Principal Investigator — Hadassah University Medical Organization
Locations (1):
- Hadassah University Medical Organization, Jerusalem, Jerusalem, Israel